CLINICAL TRIAL: NCT00644670
Title: A Multicenter, Twelve-Week Treatment, Single-Step Titration, Open-Label Study Assessing The Percentage Of Dyslipidemic High-Risk Patients Achieving LDL Cholesterol Targets With Atorvastatin Starting Doses Of 10 Mg, 20 Mg And 40 Mg.
Brief Title: A Study Of The Efficacy Of Atorvastatin For Lowering Cholesterol In High-Risk Patients With High Cholesterol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2581099
Record Dates: First submitted 2008-03-24; First posted 2008-03-27 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Previous Treatment with a Usual Maintenance Dose of a Statin (Experimental)
  Interventions: Drug: Atorvastatin
- Statin-Naive (Experimental)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — In previously treated patients, starting atorvastatin doses (oral tablets given once daily) of 20 mg (in patients with LDL-C levels between 115 and 164 mg/dL at baseline) or 40 mg (in patients with LDL-C levels between 165 and 235 mg/dL at baseline) were given for 6 weeks. If LDL-C target was achieved at Week 6, doses remained the same. If LDL-C target was not achieved at Week 6, doses were doubled.
  Arms: Previous Treatment with a Usual Maintenance Dose of a Statin
Drug: Atorvastatin — In statin-naive patients, starting atorvastatin doses (oral tablets given once daily) of 10 mg (in patients with LDL-C levels between 115 and 164 mg/dL at baseline), 20 mg (in patients with LDL-C levels between 165 and 174 mg/dL at baseline), or 40 mg (in patients with LDL-C levels between 175 and 235 mg/dL at baseline) were given for 6 weeks. If LDL-C target was achieved at Week 6, doses remained the same. If LDL-C target was not achieved at Week 6, doses were doubled.
  Arms: Statin-Naive

SUMMARY:
The purpose of the study is to evaluate the effectiveness of atorvastatin in lowering cholesterol and getting these high risk patients to their goals of LDL <115 mg/dl across starting doses of 10 mg, 20 mg, or 40 mg with one step titration.

ELIGIBILITY:
Inclusion Criteria:

* Dyslipidemia
* At a high risk for coronary heart disease

Exclusion Criteria:

* Use of higher than usual maintenance doses of statin drugs at screening
* Uncontrolled diabetes or high blood pressure
* Impaired liver function

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2003-06; Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects in entire group who achieved low-density lipoprotein cholesterol (LDL-C) target of <115 mg/dL | Week 12

SECONDARY OUTCOMES:
Mean percent change from baseline in LDL-C, high-density lipoprotein cholesterol (HDL-C), non-HDL-C (triglycerides of >200 mg/dL), total cholesterol, triglycerides, and apolipoprotein B for statin-naive patients | Weeks 6 and 12
Proportion of subjects across different LDL-C strata who achieved LDL-C target | Week 6
Proportion of diabetic subjects in entire group who achieved LDL-C target | Week 12
Proportion of subject on statin therapy at baseline who achieved LDL-C target and total cholesterol target (<190 mg/dL) | Week 12
Change from baseline in hemoglobin A1c levels | Week 12
Adverse events and laboratory test changes | Weeks 6 and 12
Proportion of subjects in entire group who achieved LDL-C target | Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (17):
- Belgium (17):
  - Pfizer Investigational Site, Antwerp
  - Pfizer Investigational Site, Brasschaat
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Edegem
  - Pfizer Investigational Site, Genk
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Gilly (charleroi)
  - Pfizer Investigational Site, La Louvière
  - Pfizer Investigational Site, Liège
  - Pfizer Investigational Site, Mechelen
  - Pfizer Investigational Site, Menen
  - Pfizer Investigational Site, Merksem
  - Pfizer Investigational Site, Mortsel
  - Pfizer Investigational Site, Roeselare
  - Pfizer Investigational Site, Seraing
  - Pfizer Investigational Site, Wilrijk
  - Pfizer Investigational Site, Wingene

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2581099&StudyName=A%20Study%20Of%20The%20Efficacy%20Of%20Lipitor%20For%20Lowering%20Cholesterol%20In%20High-Risk%20Patients%20With%20High%20Cholesterol